CLINICAL TRIAL: NCT02365129
Title: Activating Brown Adipose Tissue Through Exercise: Randomized Controlled Trial
Brief Title: Activating Brown Adipose Tissue Through Exercise
Acronym: ACTIBATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Hospital Clinico Universitario San Cecilio (Other); University Hospital Virgen de las Nieves (Other)
Responsible Party: Principal Investigator, Jonatan Ruiz Ruiz, Researcher, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI13/01393
Record Dates: First submitted 2015-02-03; First posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Obesity; Diabetes Mellitus; Metabolic Syndrome X
Keywords: BRITE adipose tissue; physical activity; Thermogenesis; Body Temperature Regulation; Energy Metabolism
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Metabolic Syndrome; Motor Activity | interventions — World Health Organization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care group (control) (No Intervention): Participants randomly assigned to the usual care (control) group will receive general advices from the exercise-training specialist about the positive effects of physical activity at the start of the study. The investigators will prepare informative pamphlets describing the benefits of physical activity that the investigators group has prepared for the Region of Andalucía (Southern Spain),http://www.juntadeandalucia.es/salud/servicios/contenidos/andaluciaessalud/docs/130/Guia_Recomendaciones_AF.pdf.
- Moderate-intensity group (Experimental): Exercise training based on recommendations for adults (WHO)
  Interventions: Other: Exercise training based on recommendations for adults (WHO)
- Vigorous-intensity group (Experimental): Exercise training based on recommendations for adults (WHO)
  Interventions: Other: Exercise training based on recommendations for adults (WHO)

INTERVENTIONS:
Other: Exercise training based on recommendations for adults (WHO) — The length of the trial will be 6 months. the total time of aerobic exercise in both moderate-intensity and vigorous-intensity groups will be 150 minutes/week, whereas the time needed to complete the resistance training exercises will be ≈15-30 minutes for both groups.
  Arms: Moderate-intensity group; Vigorous-intensity group

SUMMARY:
The energy burning capacity of brown adipose tissue makes it an attractive target for anti-obesity therapies. Sympathetic nervous system (SNS) is the classical regulator of brown adipose tissue; however, recent findings show a pool of novel brown adipose tissue activators that sidestep the need for stimulating the SNS, including cardiac natriuretic peptides. Of interest is that both SNS and non-SNS brown adipose tissue activators are sensitive to physical exercise, which opens new horizons and opportunities to study the potential effect of exercise-based therapeutic interventions. Moreover, a new protein released by exercise-stimulated skeletal muscle, irisin, seems to play a key role in the browning program of white adipose tissue. Most of the available evidence comes from animal studies, which is sometimes difficult to infer to human physiology. The overall objective of the ACTIBATE randomized controlled trial is to study the effect of long-term exercise training (6 months) on brown adipose tissue activity and quantity (primary outcomes) in young overweight and obese adults. The clinical significance of activating and recruiting brown adipose tissue on resting metabolic rate and cardiometabolic profile in humans will be determined. The investigators will also study at the molecular level the benefits of exercise on the regulation pathways in two different tissues: white adipose tissue and skeletal muscle, as well as identifying possible cross-talk between the exercising muscle and heart, and fat. Information from exercise-induced signaling on brown adipose tissue, white adipose tissue and skeletal muscle will help on identifying potential molecular therapeutic candidates.

DETAILED DESCRIPTION:
The energy burning capacity of brown adipose tissue (BAT) makes it an attractive target for antiobesity therapies. Sympathetic nervous system (SNS) is the classical regulator of BAT; however, recent findings show a pool of novel BAT activators that sidestep the need for stimulating the SNS. Of interest is that both SNS and non-SNS BAT activators are sensitive to physical exercise, which opens new horizons and opportunities to study the potential effect of exercise-based therapeutic interventions. Moreover, a new protein released by exercise-stimulated skeletal muscle, irisin, seems to play a key role in the browning program in white adipose tissue. Most of the available evidence comes from animal studies, which is sometimes difficult to infer to human physiology. To determine whether a controlled physical exercise program is able to facilitate BAT maintenance and function, stimulating pre-existing brown precursors and inducing the specific gene program to favor white-to-brown adipocyte transformation in humans is of clinical relevance.

The primary objective of the ACTIBATE randomized controlled trial (RCT) is to quantify the dose-effect of different exercise intensities, i.e. no exercise, moderate-intensity and vigorous-intensity, on BAT activity and mass (primary outcome), and on energy expenditure, thermogenic response to a test meal, shivering threshold, and cardiovascular disease risk factors, in young adults. The investigators will also obtain biopsies from white adipose tissue and skeletal muscle to analyse the expression of genes encoding proteins involved in the thermogenic machinery. The intervention groups will train 4-5 days/week (60 min per session) for a 24-week period.

With the final aim of making the exercise program transferable to society, the basis for the specific exercise dose in ACTIBATE is the physical activity recommendations for adults proposed by the World Health Organization. Since there is no information regarding the ideal exercise model to activate and recruit BAT, a major objective of ACTIBATE is to evaluate various exercise intensity levels that fall within the current public health recommendations to test whether higher intensity levels provides more benefit than the standard moderate-intensity level. ACTIBATE will combine both aerobic and resistance training.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 20-35 kg/m2.
* Not engaged in regular physical activity >20 min on >3 days/week.
* Not participating in a weight loss program.
* Stable weight over the last 3 months (body weight changes <3 kg).
* Normal electrocardiogram.
* Participants must be capable and willing to provide consent, understand exclusion criteria and accept the randomized group assignment.

Exclusion Criteria:

* History of cardiovascular disease.
* Diabetes or hypertension.
* Pregnancy, or planning to get pregnant during the study period.
* Medication for hypertension, hyperlipidemia, hyperuricemia or other illness.
* Beta blockers or benzodiazepins use.
* Smoking.
* Frequent exposure to cold temperatures (Granada is surrounded by high mountains where people can sky or do trekking).
* Taking medication for thyroid.
* Other significant medical conditions that are life-threatening or that can interfere with or be aggravated by exercise.
* Unwillingness to either complete the study requirements or to be randomized into control or training group.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in BAT mass and activity evaluated with Positron emission tomography/computed tomography (PET/CT) | Baseline and 6 month later (immediately after the interventions ends)

SECONDARY OUTCOMES:
Change from Baseline in gene expression of white adipose tissue, aliquots will be obtained by biopsies. | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in gene expression of muscle, aliquots will be obtained by biopsies. | Baseline and 6 month later (immediately after the interventions ends)
  Aliquots will be designated to gene expression, immunoblotting and morphologic studies.
Change from Baseline in resting energy expenditure measured through indirect calorimetry | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in meal Induced Thermogenesis measured through indirect calorimetry | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Cold Induced Thermogenesis measured through indirect calorimetry | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Body composition: fat mass. Using a Dual Energy X-ray Absorptiometry scan | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Body composition: lean body mass Using a Dual Energy X-ray Absorptiometry scan | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Shivering threshold: Temperature of water in a water perfuse vest connected to a chiller unit | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Thermic response to cold exposure with both subjective (Visual Analog Scales) and objective measures (skin and sublingual temperature) | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in subjective Thermic response to cold exposure: Visual Analog Scale | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Thermic response to a test meal with skin temperature | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Appetite: ad-libitum meal | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Appetite: Visual Analog Scale after a test meal | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Lipid Profile: In a blood sample | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in biomolecular markers: energy metabolism during cold exposure: In a blood sample | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Cardiorespiratory fitness measured on a maximum effort test | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Thermic response to a maximum effort test record with skin thermal receptors | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Muscular strength: 1 Repetition Maximum | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Dietary habits: 24h questionaire | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Physical activity levels: With an accelerometer | Baseline and 6 month later (immediately after the interventions ends)
Change from Baseline in Basal Heart Rate Variability: with a heart rate monitor | Baseline and 6 month later (immediately after the interventions ends)

CONTACTS AND LOCATIONS:
Overall Officials: Jonatan R Ruiz, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Granada, Spain

REFERENCES:
- [Derived] Martin-Olmedo JJ, Jurado-Fasoli L, Osuna-Prieto FJ, Garcia-Fontana C, Garcia-Fontana B, Gracia-Marco L, Munoz-Torres M, Ruiz JR. Impact of 24-week concurrent training on bone parameters and plasma levels of osteoglycin and sclerostin in young, sedentary adults: secondary analyses from the ACTIBATE randomized controlled trial. Eur J Endocrinol. 2025 Apr 30;192(5):558-567. doi: 10.1093/ejendo/lvaf087. PMID 40298018
- [Derived] Martinez-Tellez B, Xu H, Ortiz-Alvarez L, Rodriguez-Garcia C, Schonke M, Jurado-Fasoli L, Osuna-Prieto FJ, Alcantara JMA, Acosta FM, Amaro-Gahete FJ, Folkerts G, Vilchez-Vargas R, Link A, Plaza-Diaz J, Gil A, Labayen I, Fernandez-Veledo S, Rensen PCN, Ruiz JR. Effect of a 24-week supervised concurrent exercise intervention on fecal microbiota diversity and composition in young sedentary adults: The ACTIBATE randomized controlled trial. Clin Nutr. 2025 Jun;49:128-137. doi: 10.1016/j.clnu.2025.04.008. Epub 2025 Apr 15. PMID 40279809
- [Derived] Amaro-Gahete FJ, Espuch-Oliver A, Cano-Nieto A, Alcantara JMA, Garcia-Lario JV, De Haro T, Llamas-Elvira JM, Munoz Torres M, Castillo MJ, Labayen I, Ruiz JR. Impact of 24-week supervised concurrent exercise on S-Klotho and vitamin D levels: A randomized controlled trial. J Sports Sci. 2024 Dec;42(24):2562-2571. doi: 10.1080/02640414.2025.2453328. Epub 2025 Jan 20. PMID 39831661
- [Derived] Alcantara JMA, Gonzalez-Acedo A, Amaro-Gahete FJ, Plaza-Florido A. Heart Rate and Its Variability Are Associated With Resting Metabolic Rate and Substrate Oxidation in Young Women but Not in Men. Am J Hum Biol. 2024 Nov;36(11):e24157. doi: 10.1002/ajhb.24157. Epub 2024 Sep 20. PMID 39300911
- [Derived] Dote-Montero M, Acosta FM, Sanchez-Delgado G, Merchan-Ramirez E, Amaro-Gahete FJ, Labayen I, Ruiz JR. Association of meal timing with body composition and cardiometabolic risk factors in young adults. Eur J Nutr. 2023 Aug;62(5):2303-2315. doi: 10.1007/s00394-023-03141-9. Epub 2023 Apr 26. PMID 37100891
- [Derived] Jurado-Fasoli L, Di X, Sanchez-Delgado G, Yang W, Osuna-Prieto FJ, Ortiz-Alvarez L, Krekels E, Harms AC, Hankemeier T, Schonke M, Aguilera CM, Llamas-Elvira JM, Kohler I, Rensen PCN, Ruiz JR, Martinez-Tellez B. Acute and long-term exercise differently modulate plasma levels of oxylipins, endocannabinoids, and their analogues in young sedentary adults: A sub-study and secondary analyses from the ACTIBATE randomized controlled-trial. EBioMedicine. 2022 Nov;85:104313. doi: 10.1016/j.ebiom.2022.104313. Epub 2022 Oct 27. PMID 36374769
- [Derived] Ortiz-Alvarez L, Acosta FM, Xu H, Sanchez-Delgado G, Vilchez-Vargas R, Link A, Plaza-Diaz J, Llamas JM, Gil A, Labayen I, Rensen PCN, Ruiz JR, Martinez-Tellez B. Fecal microbiota composition is related to brown adipose tissue 18F-fluorodeoxyglucose uptake in young adults. J Endocrinol Invest. 2023 Mar;46(3):567-576. doi: 10.1007/s40618-022-01936-x. Epub 2022 Oct 15. PMID 36242744
- [Derived] Martinez-Tellez B, Sanchez-Delgado G, Acosta FM, Alcantara JMA, Amaro-Gahete FJ, Martinez-Avila WD, Merchan-Ramirez E, Munoz-Hernandez V, Osuna-Prieto FJ, Jurado-Fasoli L, Xu H, Ortiz-Alvarez L, Arias-Tellez MJ, Mendez-Gutierrez A, Labayen I, Ortega FB, Schonke M, Rensen PCN, Aguilera CM, Llamas-Elvira JM, Gil A, Ruiz JR. No evidence of brown adipose tissue activation after 24 weeks of supervised exercise training in young sedentary adults in the ACTIBATE randomized controlled trial. Nat Commun. 2022 Sep 12;13(1):5259. doi: 10.1038/s41467-022-32502-x. PMID 36097264
- [Derived] Merchan-Ramirez E, Sanchez-Delgado G, Arrizabalaga-Arriazu C, Acosta FM, Arias-Tellez MJ, Munoz-Torres M, Garcia-Lario JV, Llamas-Elvira JM, Ruiz JR. Circulating concentrations of free triiodothyronine are associated with central adiposity and cardiometabolic risk factors in young euthyroid adults. J Physiol Biochem. 2022 Aug;78(3):629-640. doi: 10.1007/s13105-022-00881-w. Epub 2022 Apr 6. PMID 35381950
- [Derived] Mendez-Gutierrez A, Aguilera CM, Osuna-Prieto FJ, Martinez-Tellez B, Rico Prados MC, Acosta FM, Llamas-Elvira JM, Ruiz JR, Sanchez-Delgado G. Exercise-induced changes on exerkines that might influence brown adipose tissue metabolism in young sedentary adults. Eur J Sport Sci. 2023 Apr;23(4):625-636. doi: 10.1080/17461391.2022.2040597. Epub 2022 Apr 25. PMID 35152857
- [Derived] Acosta FM, Sanchez-Delgado G, Martinez-Tellez B, Alcantara JMA, Llamas-Elvira JM, Ruiz JR. Diurnal variations of cold-induced thermogenesis in young, healthy adults: A randomized crossover trial. Clin Nutr. 2021 Oct;40(10):5311-5321. doi: 10.1016/j.clnu.2021.08.010. Epub 2021 Aug 24. PMID 34536639
- [Derived] Jurado-Fasoli L, Amaro-Gahete FJ, Merchan-Ramirez E, Labayen I, Ruiz JR. Relationships between diet and basal fat oxidation and maximal fat oxidation during exercise in sedentary adults. Nutr Metab Cardiovasc Dis. 2021 Apr 9;31(4):1087-1101. doi: 10.1016/j.numecd.2020.11.021. Epub 2020 Dec 1. PMID 33549436
- [Derived] Sanchez-Delgado G, Alcantara JMA, Acosta FM, Martinez-Tellez B, Amaro-Gahete FJ, Merchan-Ramirez E, Lof M, Labayen I, Ravussin E, Ruiz JR. Energy Expenditure and Macronutrient Oxidation in Response to an Individualized Nonshivering Cooling Protocol. Obesity (Silver Spring). 2020 Nov;28(11):2175-2183. doi: 10.1002/oby.22972. Epub 2020 Sep 27. PMID 32985119
- [Derived] Sanchez-Delgado G, Acosta FM, Martinez-Tellez B, Finlayson G, Gibbons C, Labayen I, Llamas-Elvira JM, Gil A, Blundell JE, Ruiz JR. Brown adipose tissue volume and 18F-fluorodeoxyglucose uptake are not associated with energy intake in young human adults. Am J Clin Nutr. 2020 Feb 1;111(2):329-339. doi: 10.1093/ajcn/nqz300. PMID 31826235
- [Derived] Acosta FM, Sanchez-Delgado G, Martinez-Tellez B, Migueles JH, Amaro-Gahete FJ, Rensen PCN, Llamas-Elvira JM, Blondin DP, Ruiz JR. Sleep duration and quality are not associated with brown adipose tissue volume or activity-as determined by 18F-FDG uptake, in young, sedentary adults. Sleep. 2019 Dec 24;42(12):zsz177. doi: 10.1093/sleep/zsz177. PMID 31555815
- [Derived] Amaro-Gahete FJ, Sanchez-Delgado G, Ara I, R Ruiz J. Cardiorespiratory Fitness May Influence Metabolic Inflexibility During Exercise in Obese Persons. J Clin Endocrinol Metab. 2019 Dec 1;104(12):5780-5790. doi: 10.1210/jc.2019-01225. PMID 31322652
- [Derived] Acosta FM, Martinez-Tellez B, Sanchez-Delgado G, Migueles JH, Contreras-Gomez MA, Martinez-Avila WD, Merchan-Ramirez E, Alcantara JMA, Amaro-Gahete FJ, Llamas-Elvira JM, Ruiz JR. Association of Objectively Measured Physical Activity With Brown Adipose Tissue Volume and Activity in Young Adults. J Clin Endocrinol Metab. 2019 Feb 1;104(2):223-233. doi: 10.1210/jc.2018-01312. PMID 30137350
- [Derived] Sanchez-Delgado G, Martinez-Tellez B, Olza J, Aguilera CM, Labayen I, Ortega FB, Chillon P, Fernandez-Reguera C, Alcantara JMA, Martinez-Avila WD, Munoz-Hernandez V, Acosta FM, Prados-Ruiz J, Amaro-Gahete FJ, Hidalgo-Garcia L, Rodriguez L, Ruiz YA, Ramirez-Navarro A, Muros-de Fuentes MA, Garcia-Rivero Y, Sanchez-Sanchez R, de Dios Beas Jimenez J, de Teresa C, Navarrete S, Lozano R, Brea-Gomez E, Rubio-Lopez J, Ruiz MR, Cano-Nieto A, Llamas-Elvira JM, Jimenez Rios JA, Gil A, Ruiz JR. Activating brown adipose tissue through exercise (ACTIBATE) in young adults: Rationale, design and methodology. Contemp Clin Trials. 2015 Nov;45(Pt B):416-425. doi: 10.1016/j.cct.2015.11.004. Epub 2015 Nov 3. PMID 26546068